CLINICAL TRIAL: NCT03341013
Title: A Phase 1, Randomized, Cross-over, Two-period Pilot Study Investigating Bioequivalence Between a Single Dose of Formulation 2 and Formulation 3 of MEDI0382 in Healthy Adult Subjects
Brief Title: A Pilot Study Investigating Bioequivalence Between a Single Dose of Formulation 2 and Formulation 3 of MEDI0382
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: D5670C00003
Record Dates: First submitted 2017-10-11; First posted 2017-11-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; GLP-1 receptor agonists
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): formulation 2 on Day 1 and formulation 3 on Day 10
  Interventions: Drug: MEDI0382 Formulation 2; Drug: MEDI0382 Formulation 3
- Sequence 2 (Experimental): formulation 3 on Day 1 and formulation 2 on Day 10
  Interventions: Drug: MEDI0382 Formulation 2; Drug: MEDI0382 Formulation 3

INTERVENTIONS:
Drug: MEDI0382 Formulation 2 — Sequence 1 Period 1 and Sequence 2 Period 2.
Drug: MEDI0382 Formulation 3 — Sequence 1 Period 2 and Sequence 2 Period 1

SUMMARY:
This is a randomized, open label, cross-over, two-period, pilot study in healthy adult subjects to evaluate the bioequivalence between formulation 2 and formulation 3 of MEDI0382 after a single subcutaneous (SC) dose. The study will be conducted at a single US center. Each subject will be randomized to receive a single 100 μg (or equimolar equivalent) SC dose of both formulation 2 and 3 of MEDI0382 on two different in-house periods separated by a washout period of 7 days. Formulation 3 of MEDI0382 has not been administered to humans previously. Blood samples for PK analyses of MEDI0382 concentrations will be taken predose and at 11 time points up to 48 hours after dosing (Days 3 and 12). Bedside plasma glucose levels will be monitored before meals and at bedtime during Days 1 and 10 and will be measured prior to breakfast on Days 2 and 11.

DETAILED DESCRIPTION:
This is a randomized, open label, cross-over, two-period, pilot study in healthy adult subjects to evaluate the bioequivalence between formulation 2 and formulation 3 of MEDI0382 after a single subcutaneous (SC) dose. The study will be conducted at a single US center. Each subject will be randomized to receive a single 100 μg (or equimolar equivalent) SC dose of both formulation 2 and 3 of MEDI0382 on two different in-house periods separated by a washout period of 7 days. Formulation 3 of MEDI0382 has not been administered to humans previously.

Subjects will receive the same absolute amount of MEDI0382, when dosed with either formulation 2 or formulation 3. Formulations of MEDI0382 will be administered via SC injection in the abdomen of subjects. Subjects will be in the study for a maximum of 59 days, which includes a screening period of up to 21 days. On Day 1, subjects will admitted to the clinic and will be randomized to receive formulation 2 and formulation 3 in one of two sequences; subjects randomized to sequence 1 will receive formulation 2 on Day 1 and formulation 3 on Day 10 and subjects randomized to sequence 2 will receive formulation 3 on Day 1 and formulation 2 on Day 10.

On Day 3, subjects will be discharged from the clinic and a 7-day washout period will follow. Subjects will return to the clinic on Day 10 to receive the second dose of investigational product and will remain in-house for 3 days. After discharge on Day 12, subjects will return on Day 38 for the end of study visit. Blood samples for PK analyses of MEDI0382 concentrations will be taken predose and at 11 time points up to 48 hours after dosing (Days 3 and 12). Bedside plasma glucose levels will be monitored before meals and at bedtime during Days 1 and 10 and will be measured prior to breakfast on Days 2 and 11.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects age 18 through 45 years at the time of screening.
2. Provision of signed and dated written informed consent prior to study-specific procedures.
3. Body mass index between 19 and 30 kg/m2 (inclusive) at screening
4. Good general health as judged by the investigator, based on medical history, physical examination including 12-lead ECG, vital signs, and blood and urinary laboratory assessments.
5. Female subjects of childbearing potential must have a negative pregnancy test at screening and randomization and must not be lactating.
6. Females of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception (see Section 10.2 for definition of females of childbearing potential and for a description of highly effective methods of contraception) from screening and must agree to continue using such precautions through to the end of the study. It is strongly recommended for the male partner of a female subject to also use a male condom plus spermicide throughout this period. Cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception.

Exclusion Criteria:

1. History of, or any existing condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product, put the subject at risk, influence the subject's ability to participate, or affect the interpretation of the results of the study
2. Impaired renal function, defined as s-creatinine ≥ 130 µmol/L
3. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2
4. Blood pressure and heart rate in supine position outside the ranges of 90-140 mmHg systolic, 50-90 mmHg diastolic and heart rate 40-100 beats/min following a 10-minute rest period.
5. Any clinically significant abnormal ECG, as judged by the investigator
6. Active hepatitis B, measured by positive tests of surface antigen HBsAg and/or active hepatitis C, measured by positive hepatitis C virus antibody tests
7. Positive human immunodeficiency virus antibodies
8. Known or suspected allergy to MEDI0382, any component of the formulation, or related products
9. Use of any prescription or nonprescription medication, except for paracetamol, hormonal contraceptives, and vitamins within the last 72 hours prior to check-in
10. History of alcoholism or drug abuse during the last 12 months
11. Smoking of cigarettes or other tobacco products
12. Habitual excessive consumption of methylxanthine-containing (theophylline, caffeine or theobromine) beverages and foods (coffee, tea, soft drinks such as red bull, cola, chocolate) as judged by the investigator
13. Blood donation within the last 3 months
14. Participation in any other trial investigating other products or involving blood sampling within the past 30 days
15. Potentially noncompliant or uncooperative, as judged by the investigator
16. Substance dependence likely to impact subject safety or compliance with study procedures
17. Psychiatric illness such that subjects have been committed to an institution by way of official or judicial order
18. Involvement of any AstraZeneca, MedImmune, the contract research organization, or the study site employee or their close relatives

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
Area under the drug concentration curve | 48 hours
  To evaluate bioequivalence between formulation 2 and formulation 3 of MEDI0382
Maximum observed plasma concentration of MEDI0382 | 48 hours
  To evaluate bioequivalence between formulation 2 and formulation 3 of MEDI0382.

SECONDARY OUTCOMES:
Area under the plasma drug concentration versus time curve from zero to infinity and to last observation | 48 hours
  To compare the pharmacokinetic (PK) profiles of MEDI0382 formulation 2 versus formulation 3.
Time to maximum observed plasma drug concentration | 48 hours
  To compare the pharmacokinetic (PK) profiles of MEDI0382 formulation 2 versus formulation 3.
Terminal phase elimination half-life | 48 hours
  To compare the pharmacokinetic (PK) profiles of MEDI0382 formulation 2 versus formulation 3.
Apparent clearance | 48 hours
  To compare the pharmacokinetic (PK) profiles of MEDI0382 formulation 2 versus formulation 3.
Adverse Events | 38 days
  To evaluate the safety and tolerability of a single dose of MEDI0382 in formulation 2 and 3.
12 lead electrocardiogram including RR, PR, QRS, QT, and QTc intervals | 38 days
  To evaluate the safety and tolerability of a single dose of MEDI0382 in formulation 2 and 3.
Anti-drug antibody titer | 38 days
  To evaluate the immunogenicity of a single dose of MEDI0382 in formulation 2 and 3.
Vital signs (temperature) | 38 days
  To evaluate the safety and tolerability of a single dose of MEDI0382 in formulation 2 and 3
Anti-drug antibody incidence | 38 days
  To evaluate the immunogenicity of a single dose of MEDI0382 in formulation 2 and 3.
Clinical laboratory assessments (hematology) | 38 days
  To evaluate the safety and tolerability of a single dose of MEDI0382 in formulation 2 and 3
Vital signs (systolic and diastolic blood pressure) | 38 days
  To evaluate the safety and tolerability of a single dose of MEDI0382 in formulation 2 and 3.
Vital signs (pulse rate and respiratory rate) | 38 days
  To evaluate the safety and tolerability of a single dose of MEDI0382 in formulation 2 and 3
Clinical laboratory assessments (serum chemistry) | 38 days
  To evaluate the safety and tolerability of a single dose of MEDI0382 in formulation 2 and 3
Clinical laboratory assessments (urinalysis) | 38 days
  To evaluate the safety and tolerability of a single dose of MEDI0382 in formulation 2 and 3

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Dallas, Texas, United States